CLINICAL TRIAL: NCT00446914
Title: High Blood Pressure Strategy: Hypertension Management Initiative Study
Brief Title: High Blood Pressure Strategy (HBPS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heart and Stroke Foundation of Ontario (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sheldon Tobe, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 474-2006; NCT00425828 (obsolete NCT alias)
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Systems Change (High Blood Pressure Strategy)

SUMMARY:
This program developed by the HSFO aims at helping people of Ontario and their primary healthcare providers better diagnose, manage and control high blood pressure. The High Blood Pressure Strategy brings together healthcare providers and patients to improve the way in which family doctors, nurse practitioners and pharmacists work together and with patients towards improved control of high blood pressure through the use of evidence-informed tools combined with local systems change.

DETAILED DESCRIPTION:
Approximately 5,000 patients will participate in the study at 11 family practice sites throughout Ontario. Each of the 11 clinic sites will be randomised to either intervention or delayed intervention 9 months later. The intervention is a systems change involving interprofessional education and management tools to bring together physicians, nurses and pharmacists with the patient. Patients will be monitored by their family doctor or nurse practitioner at scheduled follow-up visits during a period of 36 months for an effect of the intervention over time on the patient's blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* History of elevated BP reading or primary hypertension diagnosis

Exclusion Criteria:

* Major mental health illness of cognitive impairment
* Language barrier (unable to speak or read English)
* Lives in a long-term care home
* Secondary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon W Tobe, MD, FRCP(C), Principal Investigator — Sunnybrook Health Sciences Centre; Margaret Moy Lum-Kwong, BSc.N., MBA, CHE, Principal Investigator — Heart and Stroke Foundation of Ontario; Shirley Von Sychowski, BA, MA, Principal Investigator — Heart and Stroke Foundation of Ontario
Locations (1):
- Heart and Stroke Foundation of Ontario, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tobe SW, Moy Lum-Kwong M, Perkins N, Von Sychowski S, Sebaldt RJ, Kiss A. Heart and Stroke Foundation of Ontario (HSFO) high blood pressure strategy's hypertension management initiative study protocol. BMC Health Serv Res. 2008 Dec 10;8:251. doi: 10.1186/1472-6963-8-251. PMID 19068141